CLINICAL TRIAL: NCT03744754
Title: Fertility Preservation in Case of Endometriosis : Observational Cohort Study
Brief Title: Fertility Preservation in Case of Endometriosis
Acronym: PREFENDO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP180260
Record Dates: First submitted 2018-10-10; First posted 2018-11-16 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Endometriosis
Keywords: Fertility Preservation; Endometriosis; Endometriomas; Ovarian stimulation; Oocyte vitrification
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of follicular fluid, blood, endometrial samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with endometriosis: Women with endometriosis disease aged 18-36 years, with appropriate endometriosis diagnosis, based on transvaginal sonography, magnetic resonance imaging and/or previous surgery.Ovarian reserve was assessed by antral follicle counting (AFC) and measurement of serum anti-Mullerian hormone (AMH) levels Enrolled after preservation fertility procedure (vitrification of mature oocytes)

SUMMARY:
Fertility Preservation is now considered as crucial for the well-being of women battling cancer. However, others indications have more recently emerged. Women with endometriosis may represent a suitable group since they are at risk for compromise ovarian reserve. Data on FP in endometriosis patients are rare: only small retrospective study, case-reports and opinion publications .Nowadays, there is no available data concerning real indications for PF on endometriosis patients (endometriomas, risk of surgery, deep endometriosis?), criteria for eligibility (ovarian reserve parameters, age), quality of oocytes and number of oocytes necessary to give at least one live birth.

We propose a monocentric observational cohort study, evaluating the efficacy of oocytes cryopreservation as fertility preservation procedure, in young adult female subjects with endometriosis, to finally define the criteria of eligibility for PF procedures in case of endometriosis.

DETAILED DESCRIPTION:
Monocentric observational cohort study, enrolling young patients with endometriosis, without birth project for the moment, and asking for fertility preservation, in order to preserve mature oocytes.

Protocol of this study :

* information and signatures of consent file ;
* ovarian stimulation, oocytes retrieval and mature oocytes cryopreservation (one or more procedures)
* questionnaires every year, describing quality of life in this context of endometriosis and evolution (treatment, surgery, ART, pregnancies)
* data about number and rate of thawed oocytes after preservation, pregnancy rate and live birth rate with these oocytes.

ELIGIBILITY:
Inclusion Criteria:

* women from 18 to 36 years old
* endometriosis disease proved by sonography, MRI and/or surgery
* Consenting to participate to the study

Exclusion Criteria:

* Any contraindication for ovarian stimulation.
* Any contraindication for pregnancy .- Impossible Follow-up.

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients suffering from endometriosis, referred to our tertiary care university hospital for fertility preservation, from 18 to 36 years old.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-12-04 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
characteristics of patients who will benefit from preservation fertility in case of endometriosis (age, parameters of ovarian reserve, endometriosis stage and lesions, previous treatment or surgeries, previous fertility treatment) | 5 years
  baseline data

SECONDARY OUTCOMES:
rate of patients who will re-use their cryopreserved oocytes | 5 years
  follow up data
oocytes survival rate | 5 years
  follow up data
pregnancy rate | 5 years
  follow up data
birth rate | 5 years
  follow up data
live birth rate | 5 years
  follow up data
Quality of life, during and after preservation fertility procedure assessed by SF-36 questionnaire | 5 years
  Patients complete a SF-36 questionnaire
Events between fertility preservation and re-use or end of the study 1 | 5 years
  Nature of surgical procedures for endometriosis during the year
Events between fertility preservation and re-use or end of the study 2 | 5 years
  Number of surgical procedures for endometriosis during the year
Events between fertility preservation and re-use or end of the study 3 | 5 years
  Pregnancy during the year (and type of pregnancy: abortion, clinical pregnancy, delivery)
Events between fertility preservation and re-use or end of the study 4 | 5 years
  Duration of medical treatement for endometriosis during the year: number of months during the year
Events between fertility preservation and re-use or end of the study 5 | 5 years
  Type of medical treatement for endometriosis during the year: class of molecule

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle Mathieu d'Argent, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Gynécologie Obstétrique et Médecine de la Reproduction Hôpital TENON, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided